CLINICAL TRIAL: NCT05998993
Title: Phase II Study to Evaluate the Efficacy and Safety of SBRT as an Adjunctive Intervention for Oligoresidual Disease in EGFR Mutant NSCLC With First-Line Osimertinib Treatment
Brief Title: Study to Evaluate SBRT for EGFR Mutant NSCLC Patients Receiving Osimertinib (CULTRO)
Acronym: CULTRO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Tratamiento e Investigación sobre Cáncer, Luis Carlos Sarmiento Angulo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTIC001
Record Dates: First submitted 2023-07-28; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: EGF-R Positive Non-Small Cell Lung Cancer; Non Small Cell Lung Cancer; EGFR Exon 19 Deletion; EGFR Exon 21 Mutation; EGFR G719X
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiation (Experimental): A total of 35 patients diagnosed and treated at CTIC Centro de Tratamiento e Investigación Sobre Cáncer Luis Carlos Sarmiento Angulo.
  Interventions: Radiation: Stereotactic Body Radiation Therapy SBRT

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy SBRT — This is a non-randomized Phase II study in which all patients receive the experimental treatment with Stereotactic Ablative Radiotherapy (SABR) to residual tumor lesions (up to 5 residual metastatic lesions in a maximum of 2 organs) following 12 weeks of systemic treatment with Osimertinib. The study aims to enroll 35 patients diagnosed and treated at CTIC Centro de Tratamiento e Investigación Sobre Cáncer Luis Carlos Sarmiento Angulo.
  Other Names: Stereotactic radiosurgery SRS

SUMMARY:
Phase II Study to Evaluate the Impact of SBRT (Stereotactic Body Radiation Therapy) and/or SRS (Stereotactic Radiosurgery) on Oligoresidual Disease in EGFR Mutation Patients Treated with Osimertinib as First-Line Systemic Intervention. All candidates must exhibit a partial response after 12 weeks of treatment with the third-generation tyrosine kinase inhibitor (alone or in combination with chemotherapy) and a maximum of five (5) residual lesions in a maximum of two (2) organs. The primary outcome will be progression-free survival (PFS), and secondary outcomes will include overall survival (OS), proportion of patients without progression at months 12 and 36, safety, and overall response rate (ORR). Additionally, an exploratory analysis will be conducted on the prognostic value of liquid biopsy (supplementary information), considering baseline presence of mutations (determined by Next Generation Sequencing tests) and reduction or negativization of allelic fraction (AF).

DETAILED DESCRIPTION:
Phase II study with a single-stage Fleming design based on a normal approximation to the binomial distribution, with a one-sided type I error of 10% and a power of 90% to detect 30 events related to disease progression. Under the alternative hypothesis to detect a 35% improvement in PFS, 35 patients are required to be recruited over 22 months, with a minimum median follow-up of 14 months. An interim analysis will be conducted to determine early termination of the study using a Lan-DeMets monitoring boundary and an O'Brien-Fleming stopping rule. The interim analysis will be performed when 20 out of the expected 30 events have been observed. Employing the O'Brien-Fleming statistic, the critical value for the Z-score in the interim analysis (to stop and reject the null hypothesis) will be 1.054, and the critical value for the Z-score to stop and reject the alternative (futility) will be -0.204.

ELIGIBILITY:
Inclusion Criteria:

* Be older than 18 years of age.
* Be capable of giving informed consent to participate in the study.
* Have histological confirmation compatible with EGFR mutant non-small cell lung cancer (NSCLC) and metastatic disease (with or without histological confirmation of metastatic lesions).
* Have confirmation of the presence of common EGFR mutations (exon 19 deletion, L858R/exon 21, or G719X) through any locally and internationally accepted standard tests.
* Have received at least 12 weeks of Osimertinib treatment (with or without the addition of chemotherapy based on FLAURA2 study results after discussion with the investigative team).
* Have a partial response defined by RECIST 1.1 criteria.
* Have a maximum of 5 residual tumor lesions in up to 2 organs suitable for treatment with Stereotactic Ablative Radiotherapy (SABR).
* Have the following imaging and clinical tests within 4 weeks before study entry:
* Contrast-enhanced brain MRI.
* Chest/abdomen/pelvis CT scan, with or without bone scan (at the investigator's discretion) if PET-CT was not performed.
* 18-FDG PET-CT.
* Spinal MRI for patients with vertebral or paravertebral metastases.
* Electrocardiogram (EKG) and transthoracic echocardiogram.
* Complete blood count and standard blood chemistry.
* Negative pregnancy test for fertile women within 4 weeks prior to starting radiotherapy.
* Liquid biopsy for assessment of tumor allelic fraction (baseline).
* ECOG performance status 0-2.
* All sites of oligoresidual disease must be safely treatable according to the following criteria:
* All brain lesions must be treatable with SRS.
* The maximum size for extracranial lesions will be up to 6 cm, with exceptions for bone metastases which may include lesions larger than 6 cm at the discretion of the investigative medical team (e.g., ribs, scapula, or pelvis).
* Life expectancy >6 months.
* Not eligible for surgical treatment.
* Osimertinib treatment must be suspended 48 hours before the start of ablative therapy and cannot be initiated within 48 hours of receiving the last fraction. In patients receiving SBRT for central lung lesions, the suspension time for Osimertinib may be extended up to 5 days before and after ablative therapy.
* Patients may have previously received treatments such as radiofrequency or microwave ablation for oligoresidual lesions, but imaging must demonstrate that the lesion persists and is treatable with SABR.
* Metastatic tumor lesions that received initial treatment with radiosurgery cannot be included for SABR treatment.
* If initial treatment was conventional radiotherapy, SABR could be considered if safe to administer. In this case, the ablative therapy must be discussed by the investigative team.
* The eligibility and prognosis criteria will be reviewed by the multidisciplinary thoracic tumor board at CTIC Centro de Tratamiento e Investigación Sobre Cáncer Luis Carlos Sarmiento Angulo.

Exclusion Criteria:

* Severe comorbidities contraindicating radiation therapy.
* Bone metastases in the femur with a high risk of fracture.
* Complete response to Osimertinib treatment (no oligoresidual disease for ablative treatment).
* Inability to treat all oligoresidual lesions with ablative intent.
* History of pneumonitis or functionally limiting interstitial lung disease. It may be considered limiting if the patient is unable to perform DLCO maneuvers or if adjusted DLCO is less than 35% of predicted, PaO2 at Bogotá altitude with FiO2 21% is less than or equal to 50 mmHg.
* Clinical or radiological evidence of symptomatic spinal cord compression.
* Dominant brain metastatic disease requiring surgical management (e.g., imminent herniation or hydrocephalus).
* Candidate for a clinical trial with an experimental drug.
* Inability to receive Osimertinib with minimal adherence.
* Oligoresidual involvement in peritoneum, pleura, or bone marrow (non-measurable disease).
* Leptomeningeal involvement (presumed based on imaging findings or confirmed by cerebrospinal fluid cytology).
* Pregnant or breastfeeding women.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | Month 12
  Time from the initiation of systemic treatment (Osimertinib) to disease progression or death. This outcome is not influenced by second-line interventions and allows for the estimation of the relative efficacy of the treatment and its Hazard Ratio (HR)

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Month 12
  Proportion of patients with partial or complete response following the implementation of SBRT. This measurement does not include stable disease
Overall Survival (OS) | Month 12
  Time from diagnosis, the first day of systemic treatment, and implementation of SBRT to death from any cause or last follow-up
Progression-Free Time (PFT) | Month 12
  Time from the execution of SBRT to objective tumor progression, excluding death
Adverse Events and Safety | Month 12
  Adverse events will be graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 5 from the National Cancer Institute (NCI) US

CONTACTS AND LOCATIONS:
Overall Officials: Luis Rojas, MD, Principal Investigator — Centro de Tratamiento e Investigación sobre Cáncer, Luis Carlos Sarmiento Angulo
Locations (1):
- CTIC - Centro de Tratamiento e Investigación Sobre Cáncer Luis Carlos Sarmiento Angulo, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: Yes
The current study is intended to be published, even if prematurely terminated. The publication may encompass all or part of the following variations: online publication of a synopsis, abstract and/or presentation at a scientific conference, or publication of a complete scientific article.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 5 years
Access Criteria: Email to PI

REFERENCES:
- [Background] Planchard D, Popat S, Kerr K, Novello S, Smit EF, Faivre-Finn C, Mok TS, Reck M, Van Schil PE, Hellmann MD, Peters S; ESMO Guidelines Committee. Metastatic non-small cell lung cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2018 Oct 1;29(Suppl 4):iv192-iv237. doi: 10.1093/annonc/mdy275. No abstract available. PMID 30285222
- [Background] Wu YL, Zhou C, Liam CK, Wu G, Liu X, Zhong Z, Lu S, Cheng Y, Han B, Chen L, Huang C, Qin S, Zhu Y, Pan H, Liang H, Li E, Jiang G, How SH, Fernando MCL, Zhang Y, Xia F, Zuo Y. First-line erlotinib versus gemcitabine/cisplatin in patients with advanced EGFR mutation-positive non-small-cell lung cancer: analyses from the phase III, randomized, open-label, ENSURE study. Ann Oncol. 2015 Sep;26(9):1883-1889. doi: 10.1093/annonc/mdv270. Epub 2015 Jun 23. PMID 26105600
- [Background] Zhou C, Wu YL, Chen G, Feng J, Liu XQ, Wang C, Zhang S, Wang J, Zhou S, Ren S, Lu S, Zhang L, Hu C, Hu C, Luo Y, Chen L, Ye M, Huang J, Zhi X, Zhang Y, Xiu Q, Ma J, Zhang L, You C. Erlotinib versus chemotherapy as first-line treatment for patients with advanced EGFR mutation-positive non-small-cell lung cancer (OPTIMAL, CTONG-0802): a multicentre, open-label, randomised, phase 3 study. Lancet Oncol. 2011 Aug;12(8):735-42. doi: 10.1016/S1470-2045(11)70184-X. Epub 2011 Jul 23. PMID 21783417
- [Background] Mitsudomi T, Morita S, Yatabe Y, Negoro S, Okamoto I, Tsurutani J, Seto T, Satouchi M, Tada H, Hirashima T, Asami K, Katakami N, Takada M, Yoshioka H, Shibata K, Kudoh S, Shimizu E, Saito H, Toyooka S, Nakagawa K, Fukuoka M; West Japan Oncology Group. Gefitinib versus cisplatin plus docetaxel in patients with non-small-cell lung cancer harbouring mutations of the epidermal growth factor receptor (WJTOG3405): an open label, randomised phase 3 trial. Lancet Oncol. 2010 Feb;11(2):121-8. doi: 10.1016/S1470-2045(09)70364-X. Epub 2009 Dec 18. PMID 20022809
- [Background] Kobayashi S, Boggon TJ, Dayaram T, Janne PA, Kocher O, Meyerson M, Johnson BE, Eck MJ, Tenen DG, Halmos B. EGFR mutation and resistance of non-small-cell lung cancer to gefitinib. N Engl J Med. 2005 Feb 24;352(8):786-92. doi: 10.1056/NEJMoa044238. PMID 15728811
- [Background] Oxnard GR, Arcila ME, Sima CS, Riely GJ, Chmielecki J, Kris MG, Pao W, Ladanyi M, Miller VA. Acquired resistance to EGFR tyrosine kinase inhibitors in EGFR-mutant lung cancer: distinct natural history of patients with tumors harboring the T790M mutation. Clin Cancer Res. 2011 Mar 15;17(6):1616-22. doi: 10.1158/1078-0432.CCR-10-2692. Epub 2010 Dec 6. PMID 21135146
- [Background] Yu HA, Arcila ME, Rekhtman N, Sima CS, Zakowski MF, Pao W, Kris MG, Miller VA, Ladanyi M, Riely GJ. Analysis of tumor specimens at the time of acquired resistance to EGFR-TKI therapy in 155 patients with EGFR-mutant lung cancers. Clin Cancer Res. 2013 Apr 15;19(8):2240-7. doi: 10.1158/1078-0432.CCR-12-2246. Epub 2013 Mar 7. PMID 23470965
- [Background] Cross DA, Ashton SE, Ghiorghiu S, Eberlein C, Nebhan CA, Spitzler PJ, Orme JP, Finlay MR, Ward RA, Mellor MJ, Hughes G, Rahi A, Jacobs VN, Red Brewer M, Ichihara E, Sun J, Jin H, Ballard P, Al-Kadhimi K, Rowlinson R, Klinowska T, Richmond GH, Cantarini M, Kim DW, Ranson MR, Pao W. AZD9291, an irreversible EGFR TKI, overcomes T790M-mediated resistance to EGFR inhibitors in lung cancer. Cancer Discov. 2014 Sep;4(9):1046-61. doi: 10.1158/2159-8290.CD-14-0337. Epub 2014 Jun 3. PMID 24893891
- [Background] Wu YL, Ahn MJ, Garassino MC, Han JY, Katakami N, Kim HR, Hodge R, Kaur P, Brown AP, Ghiorghiu D, Papadimitrakopoulou VA, Mok TSK. CNS Efficacy of Osimertinib in Patients With T790M-Positive Advanced Non-Small-Cell Lung Cancer: Data From a Randomized Phase III Trial (AURA3). J Clin Oncol. 2018 Sep 10;36(26):2702-2709. doi: 10.1200/JCO.2018.77.9363. Epub 2018 Jul 30. PMID 30059262
- [Background] Goss G, Tsai CM, Shepherd FA, Bazhenova L, Lee JS, Chang GC, Crino L, Satouchi M, Chu Q, Hida T, Han JY, Juan O, Dunphy F, Nishio M, Kang JH, Majem M, Mann H, Cantarini M, Ghiorghiu S, Mitsudomi T. Osimertinib for pretreated EGFR Thr790Met-positive advanced non-small-cell lung cancer (AURA2): a multicentre, open-label, single-arm, phase 2 study. Lancet Oncol. 2016 Dec;17(12):1643-1652. doi: 10.1016/S1470-2045(16)30508-3. Epub 2016 Oct 14. PMID 27751847
- [Background] Yang JC, Ahn MJ, Kim DW, Ramalingam SS, Sequist LV, Su WC, Kim SW, Kim JH, Planchard D, Felip E, Blackhall F, Haggstrom D, Yoh K, Novello S, Gold K, Hirashima T, Lin CC, Mann H, Cantarini M, Ghiorghiu S, Janne PA. Osimertinib in Pretreated T790M-Positive Advanced Non-Small-Cell Lung Cancer: AURA Study Phase II Extension Component. J Clin Oncol. 2017 Apr 20;35(12):1288-1296. doi: 10.1200/JCO.2016.70.3223. Epub 2017 Feb 21. PMID 28221867
- [Background] Mok TS, Wu Y-L, Ahn M-J, Garassino MC, Kim HR, Ramalingam SS, Shepherd FA, He Y, Akamatsu H, Theelen WS, Lee CK, Sebastian M, Templeton A, Mann H, Marotti M, Ghiorghiu S, Papadimitrakopoulou VA; AURA3 Investigators. Osimertinib or Platinum-Pemetrexed in EGFR T790M-Positive Lung Cancer. N Engl J Med. 2017 Feb 16;376(7):629-640. doi: 10.1056/NEJMoa1612674. Epub 2016 Dec 6. PMID 27959700
- [Background] Soria JC, Ohe Y, Vansteenkiste J, Reungwetwattana T, Chewaskulyong B, Lee KH, Dechaphunkul A, Imamura F, Nogami N, Kurata T, Okamoto I, Zhou C, Cho BC, Cheng Y, Cho EK, Voon PJ, Planchard D, Su WC, Gray JE, Lee SM, Hodge R, Marotti M, Rukazenkov Y, Ramalingam SS; FLAURA Investigators. Osimertinib in Untreated EGFR-Mutated Advanced Non-Small-Cell Lung Cancer. N Engl J Med. 2018 Jan 11;378(2):113-125. doi: 10.1056/NEJMoa1713137. Epub 2017 Nov 18. PMID 29151359
- [Background] Ramalingam SS, Vansteenkiste J, Planchard D, Cho BC, Gray JE, Ohe Y, Zhou C, Reungwetwattana T, Cheng Y, Chewaskulyong B, Shah R, Cobo M, Lee KH, Cheema P, Tiseo M, John T, Lin MC, Imamura F, Kurata T, Todd A, Hodge R, Saggese M, Rukazenkov Y, Soria JC; FLAURA Investigators. Overall Survival with Osimertinib in Untreated, EGFR-Mutated Advanced NSCLC. N Engl J Med. 2020 Jan 2;382(1):41-50. doi: 10.1056/NEJMoa1913662. Epub 2019 Nov 21. PMID 31751012
- [Background] Al-Halabi H, Sayegh K, Digamurthy SR, Niemierko A, Piotrowska Z, Willers H, Sequist LV. Pattern of Failure Analysis in Metastatic EGFR-Mutant Lung Cancer Treated with Tyrosine Kinase Inhibitors to Identify Candidates for Consolidation Stereotactic Body Radiation Therapy. J Thorac Oncol. 2015 Nov;10(11):1601-7. doi: 10.1097/JTO.0000000000000648. PMID 26313684
- [Background] Patel S, Rimner A, Foster A, et al. Pattern of Failure in Metastatic EGFR-Mutant NSCLC Treated With Erlotinib: A Role for Upfront Radiation Therapy?: Metastatic Non-Small Cell Lung Cancer. International Journal of Radiation Oncology*Biology*Physics. 2014/11/15/ 2014;90(5, Supplement):S45-S46. doi:https://doi.org/10.1016/j.ijrobp.2014.08.233
- [Background] Xu Q, Zhou F, Liu H, Jiang T, Li X, Xu Y, Zhou C. Consolidative Local Ablative Therapy Improves the Survival of Patients With Synchronous Oligometastatic NSCLC Harboring EGFR Activating Mutation Treated With First-Line EGFR-TKIs. J Thorac Oncol. 2018 Sep;13(9):1383-1392. doi: 10.1016/j.jtho.2018.05.019. Epub 2018 May 29. PMID 29852232
- [Background] Barron F, Cardona AF, Corrales L, Ramirez-Tirado LA, Caballe-Perez E, Sanchez G, Flores-Estrada D, Zatarain-Barron ZL, Arrieta O; Latin American Consortium for the Study of Lung Cancer (CLICaP). Characteristics of progression to tyrosine kinase inhibitors predict overall survival in patients with advanced non-small cell lung cancer harboring an EGFR mutation. J Thorac Dis. 2018 Apr;10(4):2166-2178. doi: 10.21037/jtd.2018.03.106. PMID 29850120
- [Background] Cardona AF, Arrieta O, Zapata MI, Rojas L, Wills B, Reguart N, Karachaliou N, Carranza H, Vargas C, Otero J, Archila P, Martin C, Corrales L, Cuello M, Ortiz C, Pino LE, Rosell R, Zatarain-Barron ZL; CLICaP. Acquired Resistance to Erlotinib in EGFR Mutation-Positive Lung Adenocarcinoma among Hispanics (CLICaP). Target Oncol. 2017 Aug;12(4):513-523. doi: 10.1007/s11523-017-0497-2. PMID 28620690
- [Background] Gomez DR, Blumenschein GR Jr, Lee JJ, Hernandez M, Ye R, Camidge DR, Doebele RC, Skoulidis F, Gaspar LE, Gibbons DL, Karam JA, Kavanagh BD, Tang C, Komaki R, Louie AV, Palma DA, Tsao AS, Sepesi B, William WN, Zhang J, Shi Q, Wang XS, Swisher SG, Heymach JV. Local consolidative therapy versus maintenance therapy or observation for patients with oligometastatic non-small-cell lung cancer without progression after first-line systemic therapy: a multicentre, randomised, controlled, phase 2 study. Lancet Oncol. 2016 Dec;17(12):1672-1682. doi: 10.1016/S1470-2045(16)30532-0. Epub 2016 Oct 24. PMID 27789196
- [Background] Hu F, Xu J, Zhang B, Li C, Nie W, Gu P, Hu P, Wang H, Zhang Y, Shen Y, Wang S, Zhang X. Efficacy of Local Consolidative Therapy for Oligometastatic Lung Adenocarcinoma Patients Harboring Epidermal Growth Factor Receptor Mutations. Clin Lung Cancer. 2019 Jan;20(1):e81-e90. doi: 10.1016/j.cllc.2018.09.010. Epub 2018 Sep 24. PMID 30341018
- [Background] Gomez DR, Tang C, Zhang J, Blumenschein GR Jr, Hernandez M, Lee JJ, Ye R, Palma DA, Louie AV, Camidge DR, Doebele RC, Skoulidis F, Gaspar LE, Welsh JW, Gibbons DL, Karam JA, Kavanagh BD, Tsao AS, Sepesi B, Swisher SG, Heymach JV. Local Consolidative Therapy Vs. Maintenance Therapy or Observation for Patients With Oligometastatic Non-Small-Cell Lung Cancer: Long-Term Results of a Multi-Institutional, Phase II, Randomized Study. J Clin Oncol. 2019 Jun 20;37(18):1558-1565. doi: 10.1200/JCO.19.00201. Epub 2019 May 8. PMID 31067138
- [Background] Chan OSH, Lam KC, Li JYC, Choi FPT, Wong CYH, Chang ATY, Mo FKF, Wang K, Yeung RMW, Mok TSK. ATOM: A phase II study to assess efficacy of preemptive local ablative therapy to residual oligometastases of NSCLC after EGFR TKI. Lung Cancer. 2020 Apr;142:41-46. doi: 10.1016/j.lungcan.2020.02.002. Epub 2020 Feb 11. PMID 32088604
- [Background] Zeng Y, Ni J, Yu F, Zhou Y, Zhao Y, Li S, Guo T, Chu L, Yang X, Chu X, Cai X, Zhu Z. The value of local consolidative therapy in Osimertinib-treated non-small cell lung cancer with oligo-residual disease. Radiat Oncol. 2020 Aug 27;15(1):207. doi: 10.1186/s13014-020-01651-y. PMID 32854745
- [Background] Milano MT, Katz AW, Schell MC, Philip A, Okunieff P. Descriptive analysis of oligometastatic lesions treated with curative-intent stereotactic body radiotherapy. Int J Radiat Oncol Biol Phys. 2008 Dec 1;72(5):1516-22. doi: 10.1016/j.ijrobp.2008.03.044. Epub 2008 May 19. PMID 18495378
- [Background] Kok PS, Cho D, Yoon WH, Ritchie G, Marschner I, Lord S, Friedlander M, Simes J, Lee CK. Validation of Progression-Free Survival Rate at 6 Months and Objective Response for Estimating Overall Survival in Immune Checkpoint Inhibitor Trials: A Systematic Review and Meta-analysis. JAMA Netw Open. 2020 Sep 1;3(9):e2011809. doi: 10.1001/jamanetworkopen.2020.11809. PMID 32897371
- [Background] Prasad V, Kim C, Burotto M, Vandross A. The Strength of Association Between Surrogate End Points and Survival in Oncology: A Systematic Review of Trial-Level Meta-analyses. JAMA Intern Med. 2015 Aug;175(8):1389-98. doi: 10.1001/jamainternmed.2015.2829. PMID 26098871
- [Background] Diez P, Hanna GG, Aitken KL, van As N, Carver A, Colaco RJ, Conibear J, Dunne EM, Eaton DJ, Franks KN, Good JS, Harrow S, Hatfield P, Hawkins MA, Jain S, McDonald F, Patel R, Rackley T, Sanghera P, Tree A, Murray L. UK 2022 Consensus on Normal Tissue Dose-Volume Constraints for Oligometastatic, Primary Lung and Hepatocellular Carcinoma Stereotactic Ablative Radiotherapy. Clin Oncol (R Coll Radiol). 2022 May;34(5):288-300. doi: 10.1016/j.clon.2022.02.010. Epub 2022 Mar 7. PMID 35272913
- [Background] Hanna GG, Murray L, Patel R, Jain S, Aitken KL, Franks KN, van As N, Tree A, Hatfield P, Harrow S, McDonald F, Ahmed M, Saran FH, Webster GJ, Khoo V, Landau D, Eaton DJ, Hawkins MA. UK Consensus on Normal Tissue Dose Constraints for Stereotactic Radiotherapy. Clin Oncol (R Coll Radiol). 2018 Jan;30(1):5-14. doi: 10.1016/j.clon.2017.09.007. Epub 2017 Oct 13. PMID 29033164
- [Background] Arrieta O, Cardona AF, Martin C, Mas-Lopez L, Corrales-Rodriguez L, Bramuglia G, Castillo-Fernandez O, Meyerson M, Amieva-Rivera E, Campos-Parra AD, Carranza H, Gomez de la Torre JC, Powazniak Y, Aldaco-Sarvide F, Vargas C, Trigo M, Magallanes-Maciel M, Otero J, Sanchez-Reyes R, Cuello M. Updated Frequency of EGFR and KRAS Mutations in NonSmall-Cell Lung Cancer in Latin America: The Latin-American Consortium for the Investigation of Lung Cancer (CLICaP). J Thorac Oncol. 2015 May;10(5):838-843. doi: 10.1097/JTO.0000000000000481. PMID 25634006
- [Background] Carrot-Zhang J, Soca-Chafre G, Patterson N, Thorner AR, Nag A, Watson J, Genovese G, Rodriguez J, Gelbard MK, Corrales-Rodriguez L, Mitsuishi Y, Ha G, Campbell JD, Oxnard GR, Arrieta O, Cardona AF, Gusev A, Meyerson M. Genetic Ancestry Contributes to Somatic Mutations in Lung Cancers from Admixed Latin American Populations. Cancer Discov. 2021 Mar;11(3):591-598. doi: 10.1158/2159-8290.CD-20-1165. Epub 2020 Dec 2. PMID 33268447